CLINICAL TRIAL: NCT01640626
Title: The Impact of Health Education in Controlling Soil-transmitted Helminthiasis Among Orang Asli Schoolchildren
Brief Title: Impact of Health Education on School Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Ahmed Al-Delaimy, THE IMPACT OF HEALTH EDUCATION IN CONTROLLING SOIL-TRANSMITTED HELMINTHIASIS IN ORANG ASLI COMMUNITIES, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: University Of Malaya
Record Dates: First submitted 2012-07-11; First posted 2012-07-16 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Intestinal Helminthiasis
Keywords: Health Education; Soil-transmitted helminthiasis; Ascaris; Trichuris; Hookworm; Prevention and control
MeSH Terms: conditions — Intestinal helminthiasis; Health Education; Ancylostomiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health Education (Active Comparator): Deworming will be conducted in both schools. A health education package will be introduced to schoolchildren in the intervention school (School A) only. Both schools will be followed up for 6 months.
  Interventions: Other: Health Education package
- Control (No Intervention): Schoolchildren in school B will serve as a control group. No intervention (Health education package) will be given after complete deworming at baseline.

INTERVENTIONS:
Other: Health Education package — Health Education package that covers key health messages about the proper personal hygiene practices will be given to school children in the intervention school. The package consisted of many items such as posters, comic book, song video, competitions, drawing activities, puppet show, etc.
  Arms: Health Education

SUMMARY:
There is a sever lack in application of health education intervention for Soil Transmitted Disease (STH) in rural communities and in school children among Orang Asli in Pahang in Malaysia, and also there is a lack of information on the effect of different health education aspects on STH control in Malaysia, so the investigators think that introducing such new national educational package and for the first time in Malaysian's school will help children to make some behavior changes specially for the school children aiming to use these children as an educator agents to their families and preschool brothers and sisters, to build a base for this issue and to reduce STH intensity in these rural areas, which in turn will determine the best approach to health education intervention to be applied to other rural areas in Malaysia.

DETAILED DESCRIPTION:
The World Health Organization established that infections with STH among school¬children cause malnutrition, intellectual retardation and cognitive and educational deficits.

Although school-based intervention specifically the deworming antihelminths drugs programme were introduced into school but still Orang Asli villages in Malaysia having a high intensity and higher prevalence rate for STH, therefore the objective of this article was to review other intervention means mainly the health education intervention into school children and rural community, where most of these studies concluded that health education intervention was successful in increasing knowledge and changing some of practices among people and children which in turn decreases the prevalence and intensity of the STH. Also we think applying such intervention in Malaysia would be a benefit to change knowledge and attitude towards STH, and it will be the first research study to be applied in this field.

ELIGIBILITY:
Inclusion Criteria:

* Age:7-14
* No evidence of concomitant chronic illness such as acute respiratory tract infections, mental retardation.

Exclusion Criteria:

* Age over 15

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 317 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
1- The prevalence of intestinal parasitic infections among the Orang Asli children living in the rural areas of Pahang and Selangor will be determined. | 1-2 year
  An open-label clinical trial will be carried out to investigate the impact of health package in controlling Soil Transmitted Disease (STH) infections among Orang Asli children in rural areas of Pahang and Selangor, Malaysia. After baseline screening for the eligibility of the children, all children will be screened for STH infections.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed K. Al-Delaimy, MSc, Principal Investigator — University of Malaya; Hesham M Al-Mekhlafi, PhD, Study Chair — University of Malaya
Locations (1):
- National school of Pos Betau & NAtional school of Kuala Koyan, Kuala Lipis, Pahang, Malaysia